CLINICAL TRIAL: NCT04358679
Title: Effects of Upper Limb Ergometer on Pulmonary Function Among Patients With Spinal Cord Injury.
Brief Title: Upper Limb Ergometer on Pulmonary Function Among Patients With Spinal Cord Injury.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/00592 Somia Ilyas
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Spinal Cord Injuries
Keywords: Pulmonary Function; Spinal Cord Injury; Spirometry; Ergometer
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Treatment (Active Comparator): Conventional Treatment: Deep breathing, Assisted coughing, Sustained stretching, Splinting, Bracing and Functional mobility
  Interventions: Other: Conventional Treatment
- Upper Limb ergometer training (Experimental): Conventional Treatment + Upper Limb (UL) ergo-meter exercise
  Interventions: Other: Upper Limb ergometer training

INTERVENTIONS:
Other: Conventional Treatment — Conventional Treatment:
  * Deep breathing: 10-15 reps, twice a day (BD)
  * Assisted coughing 10-15 reps, BD
  * range of motion (ROM)+ stretching 10 reps, BD
  * Tilt table standing
  Arms: Conventional Treatment
Other: Upper Limb ergometer training — Conventional Treatment + upper limb (UL) ergometry exercise UL ergometry exercise 15 to 20 mints , 2 times ,five days per week for 6 weeks.
  Arms: Upper Limb ergometer training

SUMMARY:
Randomized Control Trial, To determine the effects of arm ergometer exercise on pulmonary function of Spinal Cord Injury.

DETAILED DESCRIPTION:
The spinal cord is a tubular structure contained nervous tissue. This acts as a transmission channel of nerve signals within the brain and spinal cord. It contains grey and white matter. The grey matter consists of cell bodies of different sensory and motor neurons and white matter consists of oriented spinal tracts.

By 2007, a prospective observational study had been conducted after a disaster occurred in Pakistan which was the most cataclysmic natural disaster in country's history as a result 73000 people were lost their lives and 126000 were harmed. There was no Spinal Cord Injury (SCI) registry existed in the country but according to different estimates 650-750 had been effected of SCI.

In United States SCI incidence mainly due to higher percentage of violence-related SCIs (18%)which is higher compared to the western Europe (8%) Australia (2%). In Pakistan the most common traumatic cause of SCI was falling from different cause followed by road traffic accident (RAT) (25.2%) and functional aerobic impairment (FAI) (8.4%). The way that SCI is associated with fantastic expenses and human sufferings , yet careful statistics of SCI are not accessible in dominant of developing countries including Pakistan.

Total lung capacities become abnormal in chronic spinal cord injury patients. Changes in chest wall compliance and decreased respiratory muscle strength leads to abnormal changes in overall lung capacities.

ELIGIBILITY:
Inclusion Criteria:

* SCI at level of upper and lower thoracic spine

Exclusion Criteria:

* Cardiovascular diseases
* Active inflammation or infection going in body
* Malignancies
* Those Individuals with have psychiatric disorders
* Any other neurological condition related to brain (stroke, parkinson's etc)
* Pressure ulcers (grade 3 and grade 4)

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Forced vital Capacity (FVC) | 6 Week
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze Forced vital Capacity in Liters
Forced Expiratory Volume in 1 second (FEV1) | 6 Week
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze Forced Expiratory Volume in 1 second FEV1 in Liters
Peak Expiratory Flow (PEF) | 6 Week
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze peak expiratory flow PEF in Liter/second.

CONTACTS AND LOCATIONS:
Overall Officials: Iqbal Tariq, MsCPPT, Principal Investigator — Riphah International University
Locations (1):
- Paraplegic Center Peshawar, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maynard FM Jr, Bracken MB, Creasey G, Ditunno JF Jr, Donovan WH, Ducker TB, Garber SL, Marino RJ, Stover SL, Tator CH, Waters RL, Wilberger JE, Young W. International Standards for Neurological and Functional Classification of Spinal Cord Injury. American Spinal Injury Association. Spinal Cord. 1997 May;35(5):266-74. doi: 10.1038/sj.sc.3100432. No abstract available. PMID 9160449
- [Background] Kirshblum SC, Burns SP, Biering-Sorensen F, Donovan W, Graves DE, Jha A, Johansen M, Jones L, Krassioukov A, Mulcahey MJ, Schmidt-Read M, Waring W. International standards for neurological classification of spinal cord injury (revised 2011). J Spinal Cord Med. 2011 Nov;34(6):535-46. doi: 10.1179/204577211X13207446293695. No abstract available. PMID 22330108
- [Background] Terson de Paleville D, Lorenz D. Compensatory muscle activation during forced respiratory tasks in individuals with chronic spinal cord injury. Respir Physiol Neurobiol. 2015 Oct;217:54-62. doi: 10.1016/j.resp.2015.07.001. Epub 2015 Jul 11. PMID 26169572
- [Background] Arsh A, Darain H, Haq ZU, Zeb A, Ali I, Ilyas SM. Epidemiology of spinal cord injuries due to bomb blast attacks, managed at paraplegic centre peshawar, pakistan: a nine years retrospective study. KMUJ: KHYBER MEDICAL UNIVERSITY JOURNAL. 2017;9(2).
- [Background] Postma K, Bussmann JB, Haisma JA, van der Woude LH, Bergen MP, Stam HJ. Predicting respiratory infection one year after inpatient rehabilitation with pulmonary function measured at discharge in persons with spinal cord injury. J Rehabil Med. 2009 Sep;41(9):729-33. doi: 10.2340/16501977-0410. PMID 19774306
- [Background] Devillard X, Rimaud D, Roche F, Calmels P. Effects of training programs for spinal cord injury. Ann Readapt Med Phys. 2007 Jul;50(6):490-8, 480-9. doi: 10.1016/j.annrmp.2007.04.013. Epub 2007 Apr 24. English, French. PMID 17482709
- [Background] Kloosterman MG, Snoek GJ, Jannink MJ. Systematic review of the effects of exercise therapy on the upper extremity of patients with spinal-cord injury. Spinal Cord. 2009 Mar;47(3):196-203. doi: 10.1038/sc.2008.113. Epub 2008 Sep 30. PMID 18825160
- [Background] Postma K, Haisma JA, de Groot S, Hopman MT, Bergen MP, Stam HJ, Bussmann JB. Changes in pulmonary function during the early years after inpatient rehabilitation in persons with spinal cord injury: a prospective cohort study. Arch Phys Med Rehabil. 2013 Aug;94(8):1540-6. doi: 10.1016/j.apmr.2013.02.006. Epub 2013 Feb 14. PMID 23416767
- [Background] Torhaug T, Brurok B, Hoff J, Helgerud J, Leivseth G. Arm Cycling Combined with Passive Leg Cycling Enhances VO2peak in Persons with Spinal Cord Injury Above the Sixth Thoracic Vertebra. Top Spinal Cord Inj Rehabil. 2018 Winter;24(1):86-95. doi: 10.1310/sci17-00029. Epub 2017 Nov 20. PMID 29434464
- [Background] DeVeau KM, Harman KA, Squair JW, Krassioukov AV, Magnuson DSK, West CR. A comparison of passive hindlimb cycling and active upper-limb exercise provides new insights into systolic dysfunction after spinal cord injury. Am J Physiol Heart Circ Physiol. 2017 Nov 1;313(5):H861-H870. doi: 10.1152/ajpheart.00046.2017. Epub 2017 Jul 14. PMID 28710067
- [Background] West CR, Currie KD, Gee C, Krassioukov AV, Borisoff J. Active-Arm Passive-Leg Exercise Improves Cardiovascular Function in Spinal Cord Injury. Am J Phys Med Rehabil. 2015 Nov;94(11):e102-6. doi: 10.1097/PHM.0000000000000358. PMID 26259052
- [Background] Zhan S, Cerny FJ, Gibbons WJ, Mador MJ, Wu YW. Development of an unsupported arm exercise test in patients with chronic obstructive pulmonary disease. J Cardiopulm Rehabil. 2006 May-Jun;26(3):180-7; discussion 188-90. doi: 10.1097/00008483-200605000-00013. PMID 16738459